CLINICAL TRIAL: NCT06418646
Title: Patients' and Caregivers' Views of Multidimensional Care in Amyotropic Lateral Sclerosis in Germany
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: ALS Association (Other); German Society of Muscle Diseases (Unknown)
Responsible Party: Sponsor
Other Study IDs: ALSpsychosoz
Record Dates: First submitted 2024-05-08; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: palliative care; caregiver burden; multidimensional care
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Caregiver Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The progressive loss of physical functioning resulting from ALS leads also to high psychosocial burden for those affected, and organizational challenges related to medical care and aids. A multidimensional and -professional care is advised in order to meet the complex requirements of this disease. In Germany, medical care structures may not fulfil these high requirements, since non-medical services such as psychological support or social counselling are not regularly included in care procedures for ALS patients. Specialised palliative care is not a standard and still commonly restricted to the last weeks of life. Additionally, it is well known that caregivers of ALS patients are highly burdened, but there is a lack of support services for them.

By means of a cross-sectional, multicentre survey, we aim to investigate patients' and caregivers' perception of medical care for ALS, provided in Germany - with particular regard to psychosocial and palliative aspects. The extent to which physical, psychological, social, spiritual, practical and informational needs are subjectively met will be assessed and correlations with mental wellbeing, subjective quality of life, attitudes towards life-sustaining measures and physician-assisted suicide, as well as caregiver burden will be examined.

Currently, study planning (questionnaires and ethical approval) is already completed and recruitment was started. The study aims to recruit 500 participants from nationwide ALS-centres. Cooperating ALS-centres will be recruited via the German Network for Motoneuron Diseases (MND-Net), of which our centre is a member. It is intended to provide data-based starting points on how care of ALS patients and their caregivers can be improved in Germany, in line with their needs.

ELIGIBILITY:
Inclusion Criteria:

* patients with at least "possible ALS" according to El-Escorial-criteria
* at least 18 years old
* no impairments of behaviour or mental performance relevant to everyday life that limits the ability to make judgments or give consent (e.g. as part of a comorbid FTD)

Exclusion Criteria:

* impairments of behaviour or mental performance relevant to everyday life that limits the ability to make judgments or give consent (e.g. as part of a comorbid FTD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Amyotrophic Lateral Sclerosis and their caregivers
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
patients' satisfaction with professional care | baseline
  patients' satisfaction with professional care for potential symptoms in the six domains physical, psychological, social, spiritual, practical and informational

SECONDARY OUTCOMES:
subjective quality of life | baseline
  McGill QoL
mental wellbeing | baseline
  HADS
caregiver burden | baseline
  CBI
attitudes towards life-sustaining measures and assisted suicide | baseline

CONTACTS AND LOCATIONS:
Overall Officials: René Günther, PD Dr., Principal Investigator — University Hospital Carl Gustav Carus at Technische Universität Dresden
Locations (1):
- University Hospital Carl Gustav Carus at Technische Universität Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request including a methodologically sound proposal for the usage of data approved by the responsible review committee, data may be shared.

REFERENCES:
- [Derived] Linse K, Weber C, Reilich P, Schoberl F, Boentert M, Petri S, Rodiger A, Posa A, Otto M, Wolf J, Zeller D, Brunkhorst R, Koch J, Hermann A, Grosskreutz J, Schroter C, Gross M, Lingor P, Machetanz G, Semmler L, Dorst J, Lule D, Ludolph A, Meyer T, Maier A, Metelmann M, Regensburger M, Winkler J, Schrank B, Kohl Z, Hagenacker T, Brakemeier S, Weyen U, Weiler M, Lorenzl S, Bublitz S, Weydt P, Grehl T, Kotterba S, Lapp HS, Freigang M, Vidovic M, Aust E, Gunther R. Patients' and caregivers' perception of multidimensional and palliative care in amyotrophic lateral sclerosis - protocol of a German multicentre study. Neurol Res Pract. 2024 Jul 4;6(1):34. doi: 10.1186/s42466-024-00328-1. PMID 38961496
- See also: Related Info — http://mnd-net.de